CLINICAL TRIAL: NCT00723411
Title: A Phase III, 3-Arm, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Investigate the Impact of Diamyd on the Progression of Diabetes in Patients Newly Diagnosed With Type 1 Diabetes Mellitus (EU)
Brief Title: A Phase III Study to Investigate the Impact of Diamyd in Patients Newly Diagnosed With Type 1 Diabetes (EU)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The primary endpoint at 15 months was not met.
Sponsor: Diamyd Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D/P3/07/4
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes; Juvenile Diabetes; Diabetes type 1; Autoimmune Diabetes; Insulin dependent Diabetes; Type 1 diabetes; Type 1 diabetes mellitus; Diamyd; rhGAD65; GAD; GAD-alum
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): This arm will receive 2 subcutaneous injections with 20 µg Diamyd on Days 1 and 30, i.e., 1 prime and 1 booster dose, followed by 2 additional single doses with Diamyd 20 µg on Days 90 and 270.
  Interventions: Drug: rhGAD65
- B (Active Comparator): This arm will receive 2 subcutaneous injections with 20 µg Diamyd on Days 1 and 30, i.e., 1 prime and 1 booster dose, followed by 2 additional single doses with placebo on Days 90 and 270.
  Interventions: Drug: rhGAD65
- C (Placebo Comparator): This arm will receive 4 injections of placebo, 1 each on Days 1, 30, 90, and 270.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhGAD65 — Diamyd (rhGAD65) 20 µg injected subcutaneously at days 1, 30, 90 and 270.
  Other Names: Diamyd; GAD65; GAD-Alum; GAD
  Arms: A
Drug: rhGAD65 — Diamyd (rhGAD65) 20 µg injected subcutaneously at days 1 and 30, followed by placebo injections at days 90 and 270.
  Other Names: Diamyd; GAD; GAD65; GAD-Alum
  Arms: B
Drug: Placebo — Placebo injected subcutaneously at days 1, 30, 90 and 270
  Arms: C

SUMMARY:
The purpose of this study is to determine whether Diamyd (rhGAD65 formulated in alum) is effective in preserving the body's own insulin producing capacity in patients recently diagnosed with type 1 diabetes.

ELIGIBILITY:
Main Inclusion Criteria:

* Male and female patients between 10 and 20 years of age
* Insulin dependent type 1 diabetes mellitus diagnosed within the previous 3 months at time of screening
* Fasting C-peptide level at time of screening above 0.1 nmol/L
* Elevated GAD65 antibodies (GADA) at time of screening

Main Exclusion Criteria:

* Treatment with immunosuppressants or any anti-diabetic medications other than insulin
* A history of certain diseases or conditions (e.g. anemia, HIV, hepatitis, epilepsy, head trauma, neurological diseases or cerebrovascular accident, alcohol or drug abuse etc)
* Treatment with any vaccine within 1 month prior to planned first Diamyd dose or planned treatment with vaccine up to 2 months after the last injection with Diamyd, excluding the influenza vaccine
* Participation in other clinical trials with a new chemical entity within the previous 3 months
* Pregnancy or planned pregnancy within 1 year after the last Diamyd dose
* Presence of associated serious disease or condition which in the opinion of the investigator makes the patient non-eligible for the study

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 334 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Meal stimulated C-peptide (area under the curve) | 15 months

SECONDARY OUTCOMES:
HbA1c | 15 months
Insulin Dose | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ludvigsson, MD, PhD, Principal Investigator — Linkoeping University
Locations (70):
- Finland (6):
  - Helsingin yliopistollinen keskussairaala, Lasten ja nuorten sairaala, Helsinki
  - Kuopion yliopistollinen sairaala, Lasten klinikka, Kuopio
  - Oulun yliopistollinen sairaala, Lasten ja nuorten klinikka, Oulu
  - Seinäjoen keskussairaala, Lastentautien poliklinikka, Seinäjoki
  - Tampereen yliopistollinen sairaala, Lasten klinikka, Tampere
  - Turun yliopistollinen keskussairaala, Lastentautien Klinikka, Turku
- France (11):
  - Medecine B, Angers
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Hôpital Pellegrin Enfants, Service d'endocrinologie pédiatrique, Bordeaux
  - Hôpital Jeanne de Flandre Sce Pédiatrie, Lille
  - CHU Timone Enfants, Service de pédiatrie multidisciplinaire, Marseille
  - CHU Montpellier Hôpital Arnaud de Villeneuve, Service de Pédiatrie 1, Montpellier
  - C.H.U.Serv.Pediatrie, Nantes
  - Hopital Robert Debré, Service d'Endocrinologie, Paris
  - Hôpital Necker, Clinique Robert Debré, Diabète de l'Enfant et de l'Adolescent,, Paris
  - CHU Rennes, Rennes
  - Hôpital des Enfants, Gastroentero-nutrition-diabétologie pédiatrique, Toulouse
- Germany (7):
  - Charité Campus Virchow Childrens Hospital, Berlin
  - DRK Kliniken Westend, Berlin
  - Hannover Kinderkrankenhaus auf der Bult, Hanover
  - Klinik und Poliklinik fȕr Kinder und Jugendliche der Universität Leipzig, Leipzig
  - Klinik fȕr Kinder- und Jugendmedizin, Mȕnchen
  - KHK Wilhelmstift, Rahlstedt
  - Universitätsklinik fȕr Kinder- und Jugendmedizin, Tȕbingen, Tȕbingen
- Italy (9):
  - Unità Operativa di Pediatria, Policlinico, Bologna
  - Struttura Complessa di Diabetologia, Ospedale S. Michele, Cagliari
  - S.S. Annunziata, Clinica Pediatrica, Chieti
  - Clinica Pediatrica, Università di Genova, Genova
  - Reparto di Pediatria, Ospedale S. Raffaele, Milan
  - Diabetologia - Dipartimento Clinica Pediatrica, Ospedale Luigi Sacco, Milan
  - Azienda Ospedaliero, Universitaria di Parma, Pediatria, Parma
  - Campus Bio-Medico, Dipartimento di Diabetologia e Endocrinologia, Roma
  - Diabetologia - Dipartimento Scienze Pediatriche, Ospedale Infantile, Regina Margherita, Torino
- Netherlands (4):
  - Meander Medisch Centrum, Lokatie Elisabeth, Amersfoort
  - Diabeter, Rotterdam
  - Orbis Medisch Centrum, Sittard-Geleen
  - Haga Ziekenhuis, Lokatie Juliana Kinderziekenhuis, The Hague
- University Medical Centre Ljubljana, Department of Pediatric Endocrinology, Ljubljana, Slovenia
- Spain (9):
  - Hospital Materno-Infantil Vall Hebrón, Barcelona
  - Hospital Materno-Infantil de Cruces, Cruces / Barakaldo
  - Hospital Materno-Infantil Ramón y Cajal, Madrid
  - Hospital Materno-Infantil La Paz, Madrid
  - Hospital Materno-Infantil Carlos Haya, Málaga
  - Hospital Materno-Infantil Vírgen del Camino, Pamplona
  - Hospital Materno-Infantil Vírgen del Rocío, Seville
  - Hospital Materno-Infantil Clínico de Valencia, Valencia
  - Hospital Materno-Infantil Miguel Servet, Zaragoza
- Sweden (20):
  - Barn- och ungdomskliniken, Lasarettet, Borås
  - Barn- och ungdomskliniken, Länssjukhuset, Gävle
  - Drottning Silvias Barnsjukhus, Barn- och ungdomssjukvården, Gothenburg
  - Barn- och ungdomskliniken, Länssjukhuset, Halmstad
  - Barn- och ungdomsmedicin, Lasarettet, Helsingborg
  - Barnkliniken, Hudiksvalls Sjukhus, Hudiksvall
  - Barn- och ungdomskliniken, Länssjukhuset Ryhov, Jönköping
  - Barn- och ungdomskliniken, Lasarettet, Kalmar
  - Barn- och ungdomskliniken, Centralsjukhuset, Karlstad
  - Barn och ungdomsmedicinska kliniken, Centralsjukhuset, Kristianstad
  - Barn- och ungdomskliniken, Universitetssjukhuset, Linköping
  - Barn- och ungdomskliniken, Universitetssjukhuset, Lund
  - Barn- och ungdomscentrum, Universitetssjukhuset MAS, Malmo
  - Barn- och ungdomskliniken, Vrinnevi sjukhus, Norrköping
  - Barn- och ungdomskliniken, Universitetssjukhuset, Örebro
  - Sachsska Barnsjukhuset, Södersjukhuset, Stockholm
  - Barn- och ungdomskliniken, NU-sjukvården/NÄL, Trollhättan
  - Barn- och ungdomskliniken, Uddevalla Sjukhus, Uddevalla
  - Barn- och ungdomskliniken, Centrallasarettet, Vaxjo
  - Barn- och ungdomskliniken, Centrallasarettet, Västerås
- United Kingdom (3):
  - Maternal & Child Health Sciences, University of Dundee, Dundee
  - Children's Admin Centre, Leicester
  - Centre for Diabetes and Metabolic Medicine (DMM), Barts and The London School of Medicine and Dentistry, London

REFERENCES:
- [Derived] Tavira B, Cheramy M, Axelsson S, Akerman L, Ludvigsson J, Casas R. Effect of simultaneous vaccination with H1N1 and GAD-alum on GAD65-induced immune response. Diabetologia. 2017 Jul;60(7):1276-1283. doi: 10.1007/s00125-017-4263-x. Epub 2017 Mar 29. PMID 28357504
- [Derived] Ludvigsson J, Cheramy M, Axelsson S, Pihl M, Akerman L, Casas R; Clinical GAD-Study Group in Sweden. GAD-treatment of children and adolescents with recent-onset type 1 diabetes preserves residual insulin secretion after 30 months. Diabetes Metab Res Rev. 2014 Jul;30(5):405-14. doi: 10.1002/dmrr.2503. PMID 24302596
- [Derived] Ludvigsson J, Krisky D, Casas R, Battelino T, Castano L, Greening J, Kordonouri O, Otonkoski T, Pozzilli P, Robert JJ, Veeze HJ, Palmer J, Samuelsson U, Elding Larsson H, Aman J, Kardell G, Neiderud Helsingborg J, Lundstrom G, Albinsson E, Carlsson A, Nordvall M, Fors H, Arvidsson CG, Edvardson S, Hanas R, Larsson K, Rathsman B, Forsgren H, Desaix H, Forsander G, Nilsson NO, Akesson CG, Keskinen P, Veijola R, Talvitie T, Raile K, Kapellen T, Burger W, Neu A, Engelsberger I, Heidtmann B, Bechtold S, Leslie D, Chiarelli F, Cicognani A, Chiumello G, Cerutti F, Zuccotti GV, Gomez Gila A, Rica I, Barrio R, Clemente M, Lopez Garcia MJ, Rodriguez M, Gonzalez I, Lopez JP, Oyarzabal M, Reeser HM, Nuboer R, Stouthart P, Bratina N, Bratanic N, de Kerdanet M, Weill J, Ser N, Barat P, Bertrand AM, Carel JC, Reynaud R, Coutant R, Baron S. GAD65 antigen therapy in recently diagnosed type 1 diabetes mellitus. N Engl J Med. 2012 Feb 2;366(5):433-42. doi: 10.1056/NEJMoa1107096. PMID 22296077